CLINICAL TRIAL: NCT02024360
Title: Center for Research in Implementation Science and Prevention (CRISP) - Community Outreach - Obesity Prevention Trial (CO-OPT)
Brief Title: Community Outreach - Obesity Prevention Trial (CO-OPT)
Acronym: CO-OPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Arthur Davidson, Director, Public Health Informatics and Epidemiiology, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AHRQ 1P01HS021138-01-03
Record Dates: First submitted 2013-12-21; First posted 2013-12-31 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Overweight; Children
Keywords: obesity; overweight; children; prevention
MeSH Terms: conditions — Obesity; Overweight | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient navigation (Experimental): Patient navigator visits home to encourage health eating, active living and parental skill building
  Interventions: Behavioral: Patient navigation

INTERVENTIONS:
Behavioral: Patient navigation — 16 session (25 hour) home-based intervention with patient navigators encouraging families to adopt healthy eating, active living and parental skill building

SUMMARY:
The purpose of this research is to investigate the effectiveness of a community health worker-based program as an adjunct to clinical services regarding childhood obesity management. This family-centered program will be delivered in the community and homes of enrolled families. The primary outcome will compare change in age-gender specific body-mass-index (BMI) z-score (zBMI) over time. All Denver Health children and families will be enrolled at study inception and receive the intervention in 1 of 5 defined 6-month stepped wedge engagements. The intervention lasts for 6 months and the time prior to engagement in the intervention will serve as the control period. Intervention construct validity will be evaluated using data on diet, activity, and fitness. The primary goal is to examine the effect of the intervention in reducing the zBMI in the index patient and secondarily on any participating family members. We will test effectiveness among demographic groups under-represented in prior studies, including very young children and Latinos. Results from this study will inform future intervention modifications and permit effect size estimation and power calculations for future randomized trials that include a community health worker-based obesity prevention and treatment program. During the course of the study, an obesity registry will be designed and implemented within an integrated safety-net healthcare system to measure primary obesity outcomes in a low-income population and conduct analyses. The community health worker will be using several new technologies (e.g., text messaging and patient relationship manager [PRM]) as an adjunct when working with an obese child and his/her family. Targeted training for clients, providers and CHW will be part of the prevention strategies implemented during the grant period, these will include motivational interviewing. All of these (i.e., obesity registry, technologies and training) will have an evaluative component.

DETAILED DESCRIPTION:
Primary Aim:

Design, conduct and evaluate a pilot community health worker (CHW) feasibility study in families with at least one overweight/obese child, targeting change in primary obesity outcomes (i.e., zBMI and health behaviors using the "5-2-1-0" targets).

1. To determine the effect of a community health worker mediated childhood obesity prevention program with families on BMI in overweight and obese (O/O) children aged 2-6 years The study sample size is selected for power to evaluate specific aim 1.a.

   1. Hypothesis: Compared to children receiving delayed-intervention, a higher proportion of O/O children in the intervention group will experience a >0.1 zBMI decrease in zBMI by -age/gender over the same 12 month period.
   2. Hypothesis: Within individual subjects, compared to their own zBMI measurements 12-24 months prior, O/O children on average will experience a decrease in the slope of their BMI trajectory of >0.1 zBMI per year after starting the intervention.
2. To determine the effect of the intervention on physical activity and eating behaviors of the index patient and their family members as summarized in "5-2-1-0" daily targets (i.e., 5 fruits and vegetables, less than 2 hours screen time, 1 hour of exercise and 0 sweetened drinks).

   a. Hypothesis: Compared to baseline measures in children receiving delayed-intervention, a higher proportion of O/O children in the intervention group will experience an improvement in "5-2-1-0" measures over the same 12 month period.
3. To determine the effect of the intervention in change in parenting skills and to evaluate the effects of the intervention on weight-related quality of life measures in the parents of O/O children 2-6 years.

   1. Hypothesis: Compared to baseline measurements, scores on a validated parenting style questionnaire will be higher at the end and 6 months after the intervention.

Secondary Aims:

1. Design and implement obesity registry functionality within an integrated safety-net healthcare system to measure primary obesity outcomes in a low-income population.

   a. What was the experience of the clinicians and administrators who used the registry program? Was it feasible and acceptable in its implementation and operations? What are areas for improvement or barriers to effective use?
2. Design, deploy and evaluate technologies (e.g., text messaging and patient relationship manager [PRM]) as an aid to CHW working with an obese child and his/her family.

   1. What was the experience of the families and patients who used the text messaging and patient relationship manager program? Was it feasible and acceptable in its implementation and operations? What are areas for improvement or barriers to effective use?
   2. What was the experience of the CHW in using the text messaging and patient relationship manager program? Was it feasible and acceptable in its implementation and operations? What are areas for improvement or barriers to effective use?
   3. What was the experience of the providers and clinicians who received and used summaries of the text messaging and patient relationship manager program? Was it feasible and acceptable in its implementation and operations? What are areas for improvement or barriers to effective use?
   4. What was the experience of the CHW in using the hand-held device for recording information in the field? Was it feasible and acceptable in its implementation and operations? What are areas for improvement or barriers to effective use?
3. Design, deliver and evaluate targeted training for clients, providers and CHW to enhance obesity clinical prevention strategies, including motivational interviewing.

   1. What was the experience of the clients, providers and CHW who were trained in obesity clinical prevention strategies? Was it feasible and acceptable in its implementation and operations? What are areas for improvement or barriers to effective use?

ELIGIBILITY:
Inclusion Criteria:

* 2-6 years old with a BMI above the 85 %ile

Exclusion Criteria:

* non-English and non-Spanish speaking, any chronic conditions

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in BMI z-score | Baseline, post intervention, 6 months post intervention
  BMI z-score will be calculated for each child at the indicated times

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Davidson, MD, MSPH, Principal Investigator — Denver Health
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yun L, Boles RE, Haemer MA, Knierim S, Dickinson LM, Mancinas H, Hambidge SJ, Davidson AJ. A randomized, home-based, childhood obesity intervention delivered by patient navigators. BMC Public Health. 2015 May 23;15:506. doi: 10.1186/s12889-015-1833-z. PMID 26002612